CLINICAL TRIAL: NCT02251522
Title: A Single Time-Point Study to Evaluate the ConforMIS iTotal® (CR) Knee Replacement System Versus Off-the-Shelf Replacement
Brief Title: A Single Time-Point Study to Evaluate the ConforMIS iTotal® (CR) Knee Versus Off-the-Shelf
Acronym: STEPS
Status: Completed | Type: Observational
Sponsor: Restor3D (Industry)
Responsible Party: Sponsor
Other Study IDs: 14-001
Record Dates: First submitted 2014-09-22; First posted 2014-09-29 (Estimated); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- ConforMIS iTotal Knee Replacement System: Patients who have had an iTotal knee replacement at least 6 months prior to testing
  Interventions: Device: ConforMIS Total Knee Replacement System
- Off-the-Shelf Knee Replacement System: Patients who have had an off-the-shelf knee replacement at least 6 months prior to testing
  Interventions: Device: Off-the-Shelf Knee Replacement System

INTERVENTIONS:
Device: ConforMIS Total Knee Replacement System — Total knee replacement system using a patient specific implant.
  Groups: ConforMIS iTotal Knee Replacement System
Device: Off-the-Shelf Knee Replacement System — Total knee replacement system not using a patient specific implant.
  Groups: Off-the-Shelf Knee Replacement System

SUMMARY:
It has been noted that patients "dramatically overestimate their functional ability early after surgery." Despite use of assistive devices increasing and functional testing scores decreasing post-surgery, the patient reported outcome scores fail to show worsening. Outcome questionnaires will be administered and functional testing will be conducted on all patients to capture these changes.

DETAILED DESCRIPTION:
The functional testing used in this study consists of tests that physical therapists use daily as objective methods to assess patients' functional status. The testing is designed to closely mimic daily activities that the patients are familiar with.

ELIGIBILITY:
Inclusion Criteria:

* Implant must be at least 6 months post-op and doing well
* Patient has had a total CR knee implant
* > 18 years of age

Exclusion Criteria:

* Simultaneous bilateral procedure occurred
* BMI > 40
* Other physical disability that requires an aid for walking or disability affecting the hips, spine, contralateral knee or other joint that limits function
* Participation in another clinical study which would confound results
* Inability to complete the protocol in the opinion of the clinical staff due to safety or other reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include a 1:1 ratio of patients enrolled into both the iTotal arm and the off-the-shelf total knee arm.
Sampling Method: Non-Probability Sample
Enrollment: 873 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Functional Outcome time differences between the two groups | at least 6 months post-op
  The study primary endpoint is to compare functional testing time between patients implanted with the iTotal implant verses the off-the-shelf implants

SECONDARY OUTCOMES:
Outcomes questionnaire- Knee Society Score | At least 6 months post op
  Comparing different patient outcome scores between the two groups
Outcomes questionnaire- KOOS | At least 6 months post op
  Comparing different patient outcome scores between the two groups
Outcomes questionnaire- Forgotten Joint Score | At least 6 months post op
  Comparing different patient outcome scores between the two groups

CONTACTS AND LOCATIONS:
Overall Officials: Robert Tait, MD, Principal Investigator — Orthopaedic Institute of Henderson; Mary O'Connor, MD, Study Chair — Yale University
Locations (16):
- United States (12):
  - Denver-Vail Orthopedics, Parker, Colorado
  - Institute for Orthopaedic Surgery & Sports Medicine, Fort Myers, Florida
  - Baptist Health South Florida, Miami, Florida
  - Coastal Orthopaedic & Sports Medicine Ctr, Port Saint Lucie, Florida
  - Bethesda Orthopedic, Bethesda, Maryland
  - Excel Orthopaedic Specialists, Woburn, Massachusetts
  - Great Lakes Bone & Joint Center, Battle Creek, Michigan
  - Lederman-Kwartowitz Center for Orthopedics and Sports Medicine, West Bloomfield, Michigan
  - Orthopaedic Institute of Henderson, Henderson, Nevada
  - St. Lawrence Health System, Potsdam, New York
  - Orthopedic Specialties of Spartanburg, Spartanburg, South Carolina
  - Advanced Orthopedics & Sports Medicine, Cypress, Texas
- Germany (4):
  - Vitos Orthopädische Klinik Kassel, Kassel
  - MedArtes, Neutraubling
  - Elblandkliniken Stiftung, Radebeul
  - Sportklinik Stuttgart, Stuttgart

IPD SHARING:
Plan to Share IPD: No